CLINICAL TRIAL: NCT05984121
Title: Which is Outstanding, Local Ozone Injection or Dextrose Prolotherapy Injection in Chronic Plantar Fasciitis?: a Randomised Controlled Study"
Brief Title: Comparison of the Effectiveness of Local Ozone Injection and Dextrose Prolotherapy Injection in Chronic Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Figen Tuncay, Physical Medicine and Rehabilitation, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEU-FTR-DG-01
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Plantar Fascitis
Keywords: Local Ozon therapy; Rehabilitation; Dextroz prolotherapy; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy control group
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomly divided into 3 groups. (They will be selected by simple random sampling using the closed envelope method). They will be divided into Group 1 (local ozon injections and exercise) and group 2 (local dextroz prolotherapy and exercise) and group 3 (exercise) Outcome evalutions in the stduy will be carried out by a researcher who is blind to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Local ozon injections (Active Comparator): Local ozone therapy consists of 95-99% oxygen, 1-5% medical ozone mixture and is obtained from medical ozone generators. Medical ozone therapy contains at least 95% oxygen and at most 5% ozone. (Bocci, Velio Alvaro. 2006)
  Interventions: Drug: Local ozon injections
- Local dextroz prolotherapy injections (Active Comparator): Hypertonic dextrose prolotherapy stimulates the cells at the injection site dehydrates, causing local tissue trauma, and increases macrophage and attracts granulocytes to that area and provides tissue healing. (Hauser, Ross and et al, 2016). Kesikburun Serdar et al. in 2022 with plantar fasciitis prolotherapy injection 3 times at 2 weeks intervals in their study "They used a 15% dextrose prolotherapy solution.
  Interventions: Drug: Local dextroz prolotherapy injections
- Exercise Group (Control Group) (Other): Patients in the exercise group were treated as in the other groups during the treatment period.
  plantar fascia stretching exercises, gastrocsoleus stretching exercises, foot intrinsic muscle strengthening exercises will be taught 2 times a day 10 times each will be asked to do so. In a systematic review by Siriphorn et al. fascia stretching exercises and gastrocsoleus stretching exercises in plantar fasciitis There is evidence that it is effective. The control group was given exercise therapy We aimed to ensure that the control group was not left untreated. in case of cold application and NSAIDs other than paracetamol will be asked not to take medication.
  Interventions: Drug: Local ozon injections; Drug: Local dextroz prolotherapy injections; Other: Exercise Group

INTERVENTIONS:
Drug: Local ozon injections — Local ozone therapy is approximately 2-3 cc of medical ozone, ozone-resistant is realised by injecting subcutaneously or intramuscularly with injectors. Local ozone injection group at 0., 2. and 4. weeks with ultrasound guided medial Firstly 1.5 cc with a 25 gauge needle into the plantar fascia insertion in the plantar region "02 lidocaine injection in a sterile way and then (according to the weeks 3 cc ozone injection of 10, 15 and 20 pyg/ml will be made respectively.
  Arms: Exercise Group (Control Group); Local ozon injections
Drug: Local dextroz prolotherapy injections — Dextrose prolotherapy injection group under ultrasound guidance at weeks 0, 2 and 4 1.5 cc 30% dextrose solution and 1.5 cc 2 lidocaine mixture with a 25 gauge needle into the medial plantar region cc 2 lidocaine mixture will be made sterile with 3 cc 15% dextrose.
  Arms: Exercise Group (Control Group); Local dextroz prolotherapy injections
Other: Exercise Group — Patients will receive a conventional therapy program consisting of exercises
  Arms: Exercise Group (Control Group)

SUMMARY:
The aim of our study was to investigate the effect of local ozone injection and dextrose prolotherapy applications on pain and foot functions to compare the efficacy and to evaluate the thickness of the plantar fascia.

DETAILED DESCRIPTION:
In this study, 60 plantar fasciitis patients aged between 18 and 75 years admitted to Kırşehir Ahi Evran University Training and Research Hospital were examined. Plantar fasciitis (PF) is a common cause of heel pain associated with gait disorders.

is one of the causes and has a significant negative impact on quality of life. The diagnosis is usually made by clinical assessment and no additional investigations are required. Treatment with non-steroidal anti-inflammatory drugs, night splints and therapeutic exercises are the first choice extracorporeal shock wave therapy and plasma-rich Minimally invasive treatments such as platelet (prp) can also be applied.Plantar dextrose prolotherapy, which is another treatment method in fasciitis, improves the ligament structure strengthens and reduces pain.In 2022, Chutumstid T et al. conducted a meta-analysis and found that dextrose prolotherapy reduces pain, increases functionality and increases plantar fascia thickness in chronic plantar fasciitis.

decreased the risk of complications. Seyam Omar et al. concluded that ozone therapy can be applied subcutaneously, periarticularly and intraarticularly. It can be preferred due to its low risk and high chance of success. is a treatment method.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, both sexes
* Pain in the plantar medial calcaneal tubercle on palpation for more than 3 months
* Accepting to participate in the study
* Heel pain, especially in the first few steps in the morning, increasing with loading during the day
* Patients with an initial VAS assessment of 4 or more on a 10 cm scale

Exclusion Criteria:

* Hyperthyroidism
* Glucose6 phosphate dehydrogenase deficiency
* Ozone allergy
* Acute metabolic disease comorbidity (acute MI, acute hyperglycaemia, diabetic ketoacidosis, acute cerebrovascular disease etc.)
* Pregnancy and breastfeeding
* Malignite
* Epilepsy
* Tipl, having a history of type 2 diabetes
* History of inflammatory rheumatic disease
* History of bleeding disorders
* Use of anticoagulants other than aspirin
* Local corticosteroid injection into the plantar fascia within the last 3 months to have a story
* ESWT treatment of the plantar fascia in the last 3 months
* To have received physiotherapy to the foot, ankle area within the last 3 months
* History of foot and ankle surgery
* Active infection at the application site (cellulitis, erysipelas, etc.)
* Allergy to dextrose
* History of peripheral neuropathy
* SI radiculopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 0. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Visual analogue scale (VAS) | 2. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Visual analogue scale (VAS) | 4. week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Visual analogue scale (VAS) | 12.week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity
Foot Function Index (FFI) | 0. week
  Foot function index; 3 subgroups as pain, disability and activity limitation consists of 23 items. The pain subscale, which contains nine items, includes the foot measures the level of pain in various situations. The inadequacy sub-scale, which contains nine items scale, on the other hand, is a scale of various functional activities depending on foot problems. determines the degree of difficulty in performing the activity. The five-item activity limitation subscale The scale assesses activity limitations due to foot problems
Foot Function Index (FFI) | 2. week
  Foot function index; 3 subgroups as pain, disability and activity limitation consists of 23 items. The pain subscale, which contains nine items, includes the foot measures the level of pain in various situations. The inadequacy sub-scale, which contains nine items scale, on the other hand, is a scale of various functional activities depending on foot problems. determines the degree of difficulty in performing the activity. The five-item activity limitation subscale The scale assesses activity limitations due to foot problems
Foot Function Index (FFI) | 4. week
  Foot function index; 3 subgroups as pain, disability and activity limitation consists of 23 items. The pain subscale, which contains nine items, includes the foot measures the level of pain in various situations. The inadequacy sub-scale, which contains nine items scale, on the other hand, is a scale of various functional activities depending on foot problems. determines the degree of difficulty in performing the activity. The five-item activity limitation subscale The scale assesses activity limitations due to foot problems
Foot Function Index (FFI) | 12.week
  Foot function index; 3 subgroups as pain, disability and activity limitation consists of 23 items. The pain subscale, which contains nine items, includes the foot measures the level of pain in various situations. The inadequacy sub-scale, which contains nine items scale, on the other hand, is a scale of various functional activities depending on foot problems. determines the degree of difficulty in performing the activity. The five-item activity limitation subscale The scale assesses activity limitations due to foot problems

SECONDARY OUTCOMES:
plantar fascia thickness measurement | 0. week
  plantar fascia thickness measurement will be performed by ultrasonography
plantar fascia thickness measurement | 12. week
  plantar fascia thickness measurement will be performed by ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No